CLINICAL TRIAL: NCT00076843
Title: Phase I Study of HTLV-I-Associated Myelopathy/Tropical Spastic Paraparesis (HAM/TSP) Using the Humanized MiK-Beta-1 Monoclonal Antibody Directed Toward the IL-2L-15R-Beta; Subunit (CD122) That Blocks IL-15 Action
Brief Title: Hu Mik-Beta-1 to Treat HTLV-1-Associated Myelopathy/Tropical Spastic Paraparesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040071; 04-N-0071
Record Dates: First submitted 2006-07-12; First posted 2004-02-04 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06-25

CONDITIONS: HTLV-1
Keywords: Interleukin-15; CD8+ T-cells; HAM/TSP; HTLV-1; HTLV-1 Associated Myelopathy; Tropical Spastic Paraparesis
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Hu-Mik-beta-1 monoclonal antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hu MiK-Beta-1

SUMMARY:
This study will examine the use of the humanized Mik-Beta-1 (Hu Mik-(SqrRoot) 1) monoclonal antibody in patients with HTLV-1-associated myelopathy/tropical spastic paraparesis (HAM/TSP). Some patients infected with the human T-lymphotropic virus type 1 (HTLV-1) virus develop HAM/TSP, a disease in which the immune response to HTLV-1 becomes directed against the person's own body in what is called an autoimmune response. Hu-Mik-Beta-1 is a genetically engineered antibody that blocks the action of a chemical produced by the body during infection or inflammation called interleukin 15 (IL-15). Blocking IL-15 may prevent the autoimmune response that results in HAM/TSP.

Patients 18 years of age and older with HAM/TSP may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, and an electrocardiogram. Participants undergo the following procedures:

1. Baseline visit(s): Repeat physical examination and blood and urine tests, as well as the following:

   * Lumbar puncture: A local anesthetic is injected to numb the skin of the lower back. A needle is inserted in the space between the bones where the cerebrospinal fluid that bathes the brain and spinal cord circulates below the spinal cord. About 4 tablespoons of fluid is collected through the needle.
   * Magnetic resonance imaging (MRI): This test uses radio waves and magnets to produce images of body tissues and organs. The patient lies on a table that slides into a metal cylinder surrounded by a strong magnetic field. During part of the scan, a contrast agent is injected to brighten the images.
   * Apheresis: This procedure is used to collect large quantities of white blood cells. Whole blood is collected through a needle in an arm vein and directed into a machine that separates it into its components by spinning. The white cells and plasma are removed and the rest of the blood (red cells and platelets) is returned to the body through the same needle.
2. Hu Mik-Beta-1 treatment: Infusions of Hu Mik-Beta-1 are given through a vein every 3 weeks for nine doses. The first treatment requires at least an overnight hospital stay; subsequent infusions are given in the outpatient clinic.
3. Blood and urine tests and a physical examination at every treatment visit and a skin test at one treatment visit.
4. Research tests at the end of the 24-week treatment period, including lumbar puncture (spinal tap), MRI scan, and apheresis.
5. After completing treatment, patients have three follow-up clinic visits for blood and urine tests, and a skin test at one follow-up visit.

DETAILED DESCRIPTION:
Objectives:

In a phase I trial we wish to determine the toxicity and provide preliminary clinical response information following the administration of humanized MiK-beta-1 (Hu MiK-Beta1), a monoclonal antibody directed toward IL-2/IL-15R Beta (CD122), in patients with HTLV-I-associated myelopathy/tropical spastic paraparesis (HAM/TSP). This antibody blocks the action of IL-15, a cytokine involved in the pathogenesis of HTLV-I associated diseases and autoimmune disorders such as rheumatoid arthritis and multiple sclerosis.

Study Population:

HAM/TSP affects about 1% of patients infected with the human T lymphotropic virus type 1 (HTLV-I), manifesting as progressive myelopathy. Several features of the immune response in HAM/TSP indicate that IL-15 may be critical to its pathogenesis. HTLV-I transactivates IL-15 and IL-15 R alpha expression through its tax protein, and supports the activation of lymphocytes in HAM/TSP, as evidenced by their spontaneous proliferation in ex vivo culture. We showed that the antibody HuMiK-Beta1 could inhibit this spontaneous lymphoproliferation. In addition, IL-15 has been shown to have a preferential positive effect on the survival of CD8+ T-cells, especially those of the memory phenotype. In HAM/TSP, an extraordinarily high frequency of tax specific CD8+ T-cells in the peripheral blood and cerebrospinal fluid is postulated to participate in the damage to the central nervous system. We have demonstrated that the addition of Hu MiK-Beta1 to ex vivo cells from HAM/TSP patients led to a marked decline in tax specific CD8+ T-cells.

Design of the Study and Outcome Parameters

In this single center, open label trial, four subjects with HAM/TSP will receive 0.5 mg/kg Hu MiK-beta1 dosed every three weeks for a total of five doses, and two subjects with HAM/TSP will receive placebo (normal saline) under the same dosing schedule. In addition, following the completion of the 0.5 mg/kg dose administration in four subjects with HAM/TSP, a dose escalation study will be performed with three subjects with HAM/TSP receiving 1.0 mg/kg of Hu MiK-beta1 at three week intervals for a total of five doses per subject, and three subjects with HAM/TSP receiving 1.5 mg/kg of Hu MiK-beta1 at three week intervals for a total of five doses per subject A Total of 10 subjects will receive study drug/placebo. We anticipate consenting up to eighteen subjects to allow for up to eight dropouts. Participants who withdraw voluntarily (not due to toxicity) after initiation of the study are considered dropouts. If this occurs prior to receiving three doses of the study medication the subjects can be replaced and should have three follow-up evaluations at four-week intervals following the last dose of the study drug. Patients who voluntarily drop out after receiving at least 3 doses of the study drug will remain in the study and continue the protocol-specific evaluations. Toxicity will be assessed using standard criteria. The clinical response will be evaluated using standardized scales including expanded disability status scale, Scripps neurologic rating scale and ambulation index. In addition, viral and immunologic outcome measures will include assays of spontaneous lymphoproliferation analysis of HTLV-I tax tetramer specific CD8+ cells, HTLV-I proviral load determination and T-cell phenotype analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be at least 18 years old.

Patients must have a diagnosis of HAM/TSP as defined by the WHO criteria, including a positive HTLV-I EIA and confirmatory pattern on Western Blot analysis. Other causes of chronic progressive myelopathy are excluded by tests for serum B12 level, Lyme disease serologies, RPR, anti-nuclear antibody (ANA), extractable nuclear antigen (ENA) screen and magnetic resonance images of brain and spinal cord.

At least 7% of each patient's peripheral blood mononuclear cell population must react with anti-CD122 immunofluorescent cell staining.

Spontaneous lymphoproliferation and HTLV-I specific cytotoxic T lymphocyte responses must be demonstrated by the patient's peripheral blood mononuclear cells in ex vivo culture.

Patients must be willing to comply with all aspects of the dosing and evaluation procedure including taking the required medications and should be willing to return for the follow-up visits.

Patients must be able to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care.

EXCLUSION CRITERIA:

EDSS greater than or equal to 7 (unable to walk beyond approximately 5 meters even with aid, essentially restructed to wheelchair).

Any contraindication to monoclonal antibody therapy, including serious adverse events related to prior monoclonal antibody therapy. Patients who have received prior antibody therapy will have pertinent medical records reviewed by the study investigator. Subjects with prior monoclonal antibody use (especially murine MiK- Beta 1) and allergy/sensitivity to murine MiK- Beta 1 are excluded.

Any vaccination within 30 days prior to study entry.

Any chronic bacterial, mycobacterial, other viral (e.g. herpes virus), fungal, parasitic or protozoal infection.

History of malignancy (active or within the previous 5 years).

History or signs of immunodeficiency

Subjects with pre-existing cardiac disease, abnormal baseline echocardiogram or significantly abnormal ECG will undergo evaluation by a cardiologist, and will be excluded if, in the opinion of the cardiologist, participation in the study would compromise the safety of the patient.

Subjects with history or laboratory evidence of thrombosis or hypercoagulable state.

Concurrent medical condition that in the opinion of the investigator would compromise the safety of the patient.

HAM/TSP patients with co-existing HTLV-I associated medical conditions, such as uveitis, alveolitis or keratoconjunctivitis sicca are not excluded unless, in the opinion of the investigator, participation in the protocol would compromise the safety of the patient. However, patients with clinically significant co-morbid neuromuscular conditions such as inflammatory myopathies and neuropathies are excluded.

Patients with cognitive impairment who are unable to provide written, informed consent.

The patient has received an investigational drug for this condition within 6 months prior to entering the study.

Contraindication to prophylactic anticoagulation with low molecular weight heparin such as history of hypersensitivity to enoxaparin, haparin, pork products, or any component of the formulation (including benzyl alcohol in multiple-dose vials); thrombocytopenia associated with a positive in vitro test for antiplatelet antibodies in the presence of enoxaparin

The patient requires concurrent therapy with other immuno-modulating agents including interferons, corticosteroids and daclizumab.

Serious illness requiring systemic treatment and /or hospitalization until the subject either completes therapy or is clinically stable (in the opinion of the investigator) on therapy for at least 14 days prior to the first dose.

Abnormal screening/baseline tests exceeding any of the limits defined below:

* Total white blood cell count less than 3000/mm(3)
* Platelet count less than 85,000/mm(3)
* INR greater than or equal to 1.5
* Serum creatinine level greater than 1.5 mg/dL
* Serum alanine transaminase or aspartate transaminase levels which are greater than two times the upper limit of normal values.
* Serum creatine kinase levels that are greater than two times the upper limit of normal values.
* Serological evidence of HIV, HTLV-II, hepatitis B or C.
* Positive pregnancy test
* Positive PPD
* Positive RPR
* Positive rheumatoid factor
* Abnormal TSH
* Abnormal B12 or folate levels
* Positive Lyme ELISA or Western Blot
* Positive lupus anticoagulant

Results of any of the following tests suggestive of an alternative diagnosis that can fully account for the clinical presentation:

* Positive RPR
* Positive rheumatoid factor
* Abnormal TSH
* Abnormal B12 or folate levels
* Positive Lyme ELISA or Western Blot
* Positive lupus screen (ANA/ENA)
* Pregnant or lactating patients
* Women who are not using an acceptable method of contraception. Acceptability of various methods of contraception will be determined by the investigator. Postmenopausal or surgically sterile women must have documentation of postmenopausal status or surgical sterility available prior to enrollment.
* Men who are not practicing adequate contraception. Acceptability of various methods of contraception will be determined by the investigator. Surgically sterile men must have documentation of surgical sterility available prior to enrollment.
* Active drug or alcohol use or dependence that in the opinion of the investigator would interfere with adherence to study requirements.
* Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental or social) that is likely to affect the patient returning for follow-up visits on schedule.
* Subjects who withdraw from this study may not re-enter. Patients who have received prior investigational therapy for HAM/TSP including daclizumab and interferon must be off the investigational therapy for 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-02-03; Primary Completion 2017-10-11 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gessain A, Gout O. Chronic myelopathy associated with human T-lymphotropic virus type I (HTLV-I). Ann Intern Med. 1992 Dec 1;117(11):933-46. doi: 10.7326/0003-4819-117-11-933. PMID 1443956
- [Background] Itoyama Y, Minato S, Kira J, Goto I, Sato H, Okochi K, Yamamoto N. Spontaneous proliferation of peripheral blood lymphocytes increased in patients with HTLV-I-associated myelopathy. Neurology. 1988 Aug;38(8):1302-7. doi: 10.1212/wnl.38.8.1302. PMID 2899862
- [Background] Jacobson S, Shida H, McFarlin DE, Fauci AS, Koenig S. Circulating CD8+ cytotoxic T lymphocytes specific for HTLV-I pX in patients with HTLV-I associated neurological disease. Nature. 1990 Nov 15;348(6298):245-8. doi: 10.1038/348245a0. PMID 2146511